CLINICAL TRIAL: NCT00859625
Title: The Impact of Active Nurse Participation on Adenoma Detection During Routine Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Harry Aslanian, Associate Professor, Yale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HIC0809004192
Record Dates: First submitted 2009-03-10; First posted 2009-03-11 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2015-01

CONDITIONS: Adenoma
Keywords: colonoscopy; adenoma detection rate
MeSH Terms: conditions — Adenoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Nurse participation during colonoscope withdrawal
  Interventions: Procedure: nurse observation during colonoscope withdrawal
- 2 (No Intervention): usual colonoscopy practice

INTERVENTIONS:
Procedure: nurse observation during colonoscope withdrawal — nurse observation during colonoscope withdrawal
  Arms: 1

SUMMARY:
Hypothesis-- Nurse observation in addition to the colonoscopist while withdrawing the colonoscope from the cecum leads to a greater adenoma detection rate.

Methods- Patients presenting for screening colonoscopy are randomized to nurse observation or usual practice. Risk factors for adenoma development and the adenoma detection rate in each group will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* performance of screening colonoscopy

Exclusion Criteria:

* history of inflammatory bowel disease, gastrointestinal bleeding

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2008-11; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Adenoma detection rate | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Harry Aslanian, MD, Principal Investigator — Yale University
Locations (1):
- Yale-New Haven Hospital, New Haven, Connecticut, United States

REFERENCES:
- [Background] Rogart JN, Siddiqui UD, Jamidar PA, Aslanian HR. Fellow involvement may increase adenoma detection rates during colonoscopy. Am J Gastroenterol. 2008 Nov;103(11):2841-6. doi: 10.1111/j.1572-0241.2008.02085.x. Epub 2008 Aug 27. PMID 18759826